CLINICAL TRIAL: NCT06193538
Title: Clinical Study on the Safety and Effectiveness of NV-A01 in the Treatment of Advanced Glioma Patients
Brief Title: The Safety and Effectiveness of NV-A01 in Glioma Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wannan Medical College (Other)
Responsible Party: Principal Investigator, Jiang Xiao-chun, Professor, First Affiliated Hospital of Wannan Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023IIT003
Record Dates: First submitted 2023-09-15; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Advanced Glioblastoma Patients

STUDY DESIGN:
Intervention Model Description: This trial is a single arm, single center IIT clinical study to evaluate the safety and efficacy of NV-A01 in patients with advanced glioblastoma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intratumoral injection of NV-A01 adenovirus (Experimental)
  Interventions: Drug: Recombinant NV-A01 adenovirus injection

INTERVENTIONS:
Drug: Recombinant NV-A01 adenovirus injection — Patients with advanced glioblastoma were intratumoral injected with NV-A01. Or the NV-A01 was injected after tumor resection.

SUMMARY:
The goal of this clinical trial is to learn about the safety and effectiveness of NV-A01 in the treatment of advanced glioma patients. The main questions it aims to answer are:

1. The safety of NV-A01 in the treatment of advanced glioblastoma patients.
2. The effectiveness of NV-A01 in treating patients with advanced glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced malignant glioma confirmed by histopathology;
2. Patients who have received radiotherapy and/or temozolomide (TMZ) treatment and have residual or recurrent tumors;
3. Patients diagnosed with lesions ≥ 1.0 cm after qualified assessment;
4. KPS score ≥ 60 points;
5. The subjects had informed consent to this study before the experiment and voluntarily signed an informed consent form.

Exclusion Criteria:

1. Patients with unstable central nervous system metastases or meningeal metastases with clinical symptoms, with a risk of brain herniation or severe brain herniation, and judged by researchers as unsuitable for inclusion;
2. Patients with severe cardiovascular diseases, active autoimmune diseases, and other diseases that have been determined by researchers to be unsuitable for enrollment;
3. Patients who have received immunotherapy in the past and have an irAE level ≥ 3, and have been determined by the researchers to be unsuitable for enrollment;
4. Patients with an expected survival period of less than 3 months and judged by the researchers as unsuitable for enrollment;
5. Researchers believe that patients with other serious systemic diseases or other reasons are not suitable for participating in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerabilityof NV-A01 in the treatment of advanced glioma patients as measured by Frequency of Grade 3 or Above Adverse Events | One months after the last injection
  All events with a Grade 3 or above toxicity (defined by the NCI-CTCAE 5.0) will be tabulated by event and by relationship to NV-A01.

SECONDARY OUTCOMES:
Evaluate the effectiveness of NV-A01 in treating patients with advanced glioblastoma | Six months after the last injection
  Evaluate objective response rate (ORR), disease control rate (DCR), and progression free survival (PFS) according to the evaluation criteria for solid tumor efficacy (RECIST 1.1).
Developing pharmacodynamic indicators Discovering pharmacodynamic indicators Discovering pharmacodynamic indicators | Six months after the last injection
  Proportion of CD3+, CD4+, CD8+T cells and the expression of CD69 on the surface of T cells in peripheral blood are detected by flow cytometry. The concentration of IL2 and IFN-gamma in plasma are measured by ELISA. Samples are collected prior to the administration of NV-A01 and at regular intervals after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Chun Jiang, Doctor, Principal Investigator — Wannan Medical College Hospital
Locations (1):
- Wannan medical college hospital, Wuhu, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided